CLINICAL TRIAL: NCT00581295
Title: Use of Diffuse Optical Spectroscopy for Evaluation of the Trauma/Critically Care Patients
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Michael E. Lekawa, MD Chief, Division of Trauma/Critical Care Surgery, University of California, Irvine
Other Study IDs: 20139435
Record Dates: First submitted 2007-12-19; First posted 2007-12-27 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Trauma
Keywords: internal bleeding; changes in tissue perfusion
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- trauma: Diffuse optical spectroscopy measurment
  Interventions: Device: Diffuse optical spectroscopy

INTERVENTIONS:
Device: Diffuse optical spectroscopy — Diffuse optical spectroscopy measurment

SUMMARY:
Trauma remains the leading cause of death and disability for Americans age 1-44. Trauma can cause internal bleeding, and this bleeding is often hard to detect without sophisticate tests that take time to complete and analyze.

In addition, internal bleeding, including bleeding into the lung and chest cavity, as well as other blood loss, happens in many critically ill patients. For example, for hemorrhage, it is very difficult to detect active hemorrhage and to determine optimal rates of fluid and blood resuscitation.

Diffuse optical spectroscopy has the potential to accurately assess adequacy of tissue perfusion, oxygenation, tissue oxygen extraction, and cytochrome oxidation states that may be critical to optimal treatment, end- organ preservation, and survival.

DETAILED DESCRIPTION:
The research' want to monitor tissue perfusion and indicators of tissue damage and viability in critically ill patients by using DOS.

Non-invasive Optical Techniques DOS,near-infrared diffuse optical spectroscopy (NIR-DOS.

NIR-DOS provides functional physiologic tissue/organ information without ionizing radiation and without withdrawing any blood, in a cost-effective and rapid manner. The application of frequency-domain photon migration analysis (FDPM) to NIRS allows independent measurements of tissue absorption and scattering properties at depths of 1 cm or more below the skin surface.

Such capabilities will improve early diagnosis, detection, optimization of therapy, assessment of adequacy of resuscitation, and alteration in management plans for all of these critical conditions.

ELIGIBILITY:
Inclusion Criteria:

* Adult age 18 years or older, male or female
* Trauma/Critical Care patient

Exclusion Criteria:

* Subject is not Trauma/Critical Care patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Trauma/Critically Care Patients
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2007-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The ability to noninvasively diagnose conditions in the intensive care unit, or in battlefield conditions. | 5 to 60 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Lekawa, M.D, Principal Investigator — Beckman Laser Institute
Locations (2):
- United States (2):
  - Beckman Laser Institute,University of California, Irvine, Irvine, California
  - Trauma/Critical Care Units, UCI Medical Center, Orange, California